CLINICAL TRIAL: NCT00146497
Title: Cytokine Change in Bronchoalveolar Lavage Fluid After Early Budesonide-Surfactant Treatment in Premature Infants
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DMR92-IRB-127
Record Dates: First submitted 2005-09-04; First posted 2005-09-07 (Estimated); Last update posted 2006-06-27 (Estimated); Status verified 2006-06

CONDITIONS: Premature Infants; Respiratory Distress Syndrome; Chronic Lung Disease; Bronchoalveolar Lavage Fluid; Cytokines
Keywords: Respiratory distress syndrome (RDS); Premature infants; Chronic lung disease (CLD); Bronchoalveolar lavage fluid (BALF); Cytokines
MeSH Terms: conditions — Premature Birth; Respiratory Distress Syndrome

INTERVENTIONS:
Drug: Budesonide-Surfactant

SUMMARY:
Pulmonary inflammation plays an important role in the development of chronic lung disease (CLD) in preterm infants. This inflammation occurs very early in postnatal life. Any therapy that could be beneficial in preventing CLD should be started very early. The investigators' previous double-blind study has shown that early (< 12 hours) postnatal use of intravenous dexamethasone for 4 weeks significantly suppressed pulmonary inflammation and significantly reduced the incidence of CLD. However, the use of dexamethasone was associated with increased incidence of infection and sepsis. Their follow-up study also suggested an increase in the incidence of psychomotor anomalies. As compared to intravenous administration, endotracheal instillation will provide more local anti-inflammatory effects and less systemic side effects. Infants will be eligible for the study if their birth weight (BW) is < 1500 gm and if they had severe respiratory distress syndrome (RDS) requiring mechanical ventilation shortly after birth. After informed consent is obtained, the infant will be randomly assigned depending on the condition of the infant. The primary outcome is the change in cytokines (interleukin-6, 8, 10 and TNF-α) levels in BAL fluid. Chronic lung disease (CLD) was judged at 36 postmenstrual weeks. Infants in the study group (S/B group) received surfactant (Survanta®, Abbott Laboratories, North Chicago, IL; 100 mg or 4 mL/kg/dose) and Budesonide (Pulmicort®, AstraZeneca Pty Ltd., Australia; 0.5 mg or 1mL/kg/dose), while those in the control group (S group) received surfactant (Survanta® Abbott, 100 mg/kg/dose) and saline (1mL/kg).

DETAILED DESCRIPTION:
Growing evidence suggests that early, postnatal pulmonary inflammation may play an important role in the development of chronic lung disease (CLD) in preterm infants on mechanical ventilation.The investigator's previous study demonstrated that interleukin-8 (IL-8), a marker of inflammation, in bronchoalveolar lavage (BAL) fluid increased by as early as 2 days of age in infants who subsequently developed CLD compared with infants who did not develop the disease. Thus for any therapy to be beneficial in preventing CLD, it should be started very early. Early postnatal use of intravenous dexamethasone therapy for 4 weeks significantly suppressed pulmonary inflammation and significantly reduced the incidence of CLD. However, the use of dexamethasone was associated with increased incidence of infection and sepsis which affected the immediate outcome and contributed significantly to mortality. It was shown that school age children who had received early postnatal dexamethasone therapy for the prevention of CLD showed a significant increase in incidence of neuromotor and cognitive delay. Based on the results of these studies, early systemic dexamethasone therapy should not be recommended. Budesonide has high local anti-inflammatory activity and is one of the most extensively used inhaled glucocorticoids. Budesonide decreases airway hyperresponsiveness and reduces the number of inflammatory cells and mediators present in the airways of patients with asthma. A previous study indicated that the addition of Budesonide to Survanta did not affect the surface tension. We proposed a randomized controlled trial to study whether early endotracheal instillation of Surfactant-Budesonide (S/B) mixture would reduce lung inflammation and improve pulmonary outcome. We will measure the cytokines levels in BAL fluid to evaluate the local anti-inflammatory effect of S/B treatment.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with birth weight between 500-1500 gm
* Have severe radiographic RDS and require mechanical ventilation within 4 hours after birth

Exclusion Criteria:

* Presence of prenatal infection, congenital anomalies and lethal cardio-pulmonary status.

Ages: 1 Hour to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30
Dates: Start 2004-08

PRIMARY OUTCOMES:
The primary outcome variables are the levels of proinflammatory cytokines IL-6, IL-8 and TNF-α and anti-inflammatory cytokine IL-10.

SECONDARY OUTCOMES:
The secondary outcome is the clinical endpoint of survival free of oxygen dependence at 36 wks postmenstrual age.

CONTACTS AND LOCATIONS:
Overall Officials: Tsu-Fuh Yeh, MD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan